CLINICAL TRIAL: NCT04788147
Title: Performance and Safety of Biology-Guided Radiotherapy Using the RefleXion Medical Radiotherapy System (BIOGUIDE-X)
Acronym: BIOGUIDE-X
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RefleXion Medical (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: 985-00001
Record Dates: First submitted 2021-03-04; First posted 2021-03-09 (Actual); Results first posted 2023-10-24 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Cancer; Tumor, Solid; Cancer, Lung; Cancer, Bone; Metastasis to Lung; Metastasis to Bone
Keywords: Radiation Oncology; Radiotherapy; Biology-Guided Radiotherapy (BgRT); RefleXion Medical; Radiation Therapy
MeSH Terms: conditions — Neoplasms; Lung Neoplasms; Bone Neoplasms

STUDY DESIGN:
Intervention Model Description: This is an open-label, prospective study. The study is divided into two sequential cohorts of patients with one targetable primary or metastatic lesion in either the lungs or bone. Patients with multiple metastases can be accrued, but these investigations will focus on only one lesion per patient.
  Cohort I seeks to identify the Recommended RefleXion FDG dose (RRFD), which is the dose of administered FDG that allows for functioning of the RefleXion system. To that end, dose levels of 15 mCi and 20 mCi (if required) are assessed sequentially in an escalation protocol.
  The RRFD identified in Cohort I is utilized in Cohort II, to emulate and assess the dose delivery performance of the end-to-end BgRT workflow.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Cohort I: RRFD Cohort (Experimental): Cohort I seeks to identify the Recommended RefleXion FDG dose (RRFD), which is the dose of administered FDG that allows for functioning of the RefleXion system. This phase of the investigation seeks to optimize the balance between minimizing patient exposure to the radiotracer and achieving satisfactory performance of the RMRS PET subsystem for BgRT. The dose levels of 15 mCi and 20 mCi (if required) will be assessed sequentially in an escalation protocol. To determine the RRFD, a modified 3+3 design will be utilized wherein meeting the Activity Concentration threshold - not dose-limiting toxicity as is typically used - will be the relevant criteria for escalating from one dose to the next. Up to 12 participants will be enrolled in Cohort I, and will undergo one RMRS imaging session and one third-party Positron Emission Tomography (PET) /CT imaging session.
  Interventions: Device: RMRS IDE Device
- Cohort II: Emulated Delivery Cohort (Experimental): After the RRFD is determined by Cohort I, Cohort II enrollment will start enrollment. Cohort II seeks to determine whether BgRT dose distributions generated from Limited Time Sample (LTS) RMRS PET images obtained at the time of treatment delivery are consistent with the approved BgRT plan. To achieve this objective, RMRS PET scans will be added to the SBRT workflow at timepoints representing some of the instances when the RMRS PET subsystem would be utilized during a BgRT workflow. Specifically, subjects will undergo RMRS PET collections at the time of planning, and then before the first and final fractions of their planned course of SBRT treatment.
  Up to 22 participants will be enrolled in Cohort II, and will undergo three RMRS imaging sessions and one third-party Positron Emission Tomography (PET) /CT imaging session.
  Interventions: Device: RMRS IDE Device

INTERVENTIONS:
Device: RMRS IDE Device — Participants will be injected with FDG at the studied dose and will undergo imaging sessions using the RMRS IDE device and a third-party Positron Emission Tomography (PET)/CT imaging device.
  Other Names: RefleXion Medical; Biology-Guided Radiotherapy (BgRT)

SUMMARY:
The purpose of this study is to assess the performance and safety of Biology-Guided Radiotherapy (BgRT) using the RefleXion Medical Radiotherapy System (RMRS) via optimizing F18-Fluorodeoxyglucose (FDG) dosing, assessing the performance of the Positron Emission Tomography (PET) imaging subsystem for BgRT treatment planning and delivery, including its role as an interlock, and validating the dose delivery performance of the end-to-end BgRT workflow.

DETAILED DESCRIPTION:
The performance and safety of BgRT using the RMRS will be studied by to sequential cohorts of patients with one targetable metastatic lesion in either the lungs or bone. Patients with multiple metastases can be accrued, but these investigations will focus on only one lesion per patient.

Cohort I will seek to identify the Recommended RefleXion FDG dose (RRFD), which is the dose of administered FDG - within a range concordant with the American College of Radiology and Society of Pediatric Radiology Practice Parameter for Performing PET/CT in Oncology (ACR-SPR Practice Parameter) - that allows for functioning of the RefleXion system. Keeping ALARA ("As Low As Reasonable Achievable") principles in mind, this phase of the investigation seeks to optimize the balance between minimizing patient exposure to the radiotracer and achieving satisfactory performance of the RMRS PET subsystem for BgRT. This cohort will also seek to assess RMRS PET imaging performance in comparison to a third-party diagnostic PET/CT.

To that end, dose levels of 15 mCi and 20 mCi (if required) will be assessed sequentially in an escalation protocol. Patients with at least one known FDG avid tumor in the bone or lung will be enrolled into this cohort. These patients will undergo a CT simulation in an acceptable radiotherapy treatment position and with immobilization devices as needed. After acquisition of CT images, contours for targets, OARs, and BTZ will be generated by the investigator. Next, the patient will undergo back-to-back PET scans on the RefleXion device and a third-party diagnostic PET/CT device after a single injection of FDG at the studied FDG dose level. Quantitative metrics will be collected for each lesion in order to assess the performance of the RMRS PET subsystem at that dose. Up to 12 participant will be enrolled in Cohort I. Actual delivery of radiotherapy to the patient is not part of this investigation.

The chief objective of Cohort II is to confirm that the machine-deliverable fluence generated by applying the BgRT firing filter to PET LTS images obtained at the time of a radiotherapy delivery does in fact result in an anatomic dose distribution that is consistent with the approved BgRT plan. A secondary objective is to extend this analysis by also confirming that the linear accelerator subsystem hardware is able to deliver the received machine instructions. Importantly, this investigation comprehensively emulates and assesses (without actually delivering the radiation therapy to the patient) the entire end-to-end BgRT workflow from simulation to treatment planning to, finally, dose delivery. This design also provides an opportunity to assess imaging, workflow, and the toxicity, if any, associated with multiple administrations of FDG.

To do this, up to 22 subjects dispositioned to undergo conventional SBRT for a single bone tumor or a single lung tumor will be enrolled. As noted previously, patients with multiple metastases can be accrued but the investigation will focus only one targeted lesion per patient. For each patient, RMRS PET collections will be added to the SBRT workflow at 3 timepoints representing the steps when the RMRS PET subsystem would be utilized during the BgRT workflow. Specifically, these timepoints will include a RMRS PET imaging-only session prior to the start of SBRT delivery that will be used to create a BgRT plan as well as RMRS PET collections before the first and final fractions of their planned course of SBRT. A single comparison third-party diagnostic PET/CT image will also be obtained on the day of the final fraction.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than 21 years
2. A new or prior diagnosis of biopsy-proven cancer with a solid tumor (non-hematologic, non-lymphoma)
3. At least one active tumor in the bone or lung which is either the primary tumor or metastatic lesion determined either by biopsy or imaging suspicious of active disease
4. Target tumor size ≥2cm and ≤5cm
5. Target lesion in the bone or lung that is discrete and assessed by the investigator to be FDG-avid (i.e. SUVmax≥6 on third-party diagnostic PET/CT performed within 60 days with no intervening oncologic therapies)
6. ECOG Performance Status 0-3
7. Must have completed any other oncologic therapies at least 15 days prior to planned start of study procedures (preferably 30 days) and must have no plans to initiate systemic therapy until after study follow up is complete -OR- must be recorded by physician to have an active candidate lesion that is unresponsive to ongoing systemic therapy.
8. Females of childbearing potential should have negative urine or serum pregnancy test within 14 days prior to initiation of study scans.
9. Demonstrate adequate organ function: determined by ANC, platelets, hemoglobin, with no gross hematuria
10. For Cohort II only: Patient is dispositioned to undergo SBRT to a bone or lung tumor

Exclusion Criteria:

1. Clinically significant blood glucose abnormalities that preclude a satisfactory FDG PET/CT scan.
2. Previous history of external radiotherapy where prior radiotherapy fields are anticipated to overlap with the radiotherapy fields required for the present study
3. Diffuse metastatic process (leptomeningeal disease, peritoneal carcinomatosis, diffuse bone marrow involvement, etc.)
4. PET-avid structures not intended for radiation are within 2cm from target on third-party diagnostic PET/CT as assessed by investigator
5. Known allergy to FDG
6. Known psychiatric or substance abuse disorder that would interfere with conduct of the study
7. Pregnant, breast-feeding or expecting to conceive during the study
8. Patient weight exceeding the weight limit outlined per IFU.
9. For Cohort II only: Patients with pacemakers and other implantable devices who are deemed to be at high risk by the treating physician for complications secondary to radiotherapy.
10. For Cohort II only: Patients with bone lesions who are determined to be high risk by the treating physician for pathologic fracture prior to beginning radiotherapy.
11. For Cohort II only: Active inflammatory bowel disease, scleroderma, or other disorder deemed to be a risk factor for excess toxicity in the area of treatment by the treating physician.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-03-26 (Actual); Primary Completion 2021-12-20 (Actual); Study Completion 2021-12-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Chang, MD, Principal Investigator — Stanford University; Aurelie Garant, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (2):
- United States (2):
  - Stanford University, Stanford, California
  - UT Southwestern, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort I: Recommended RefleXion FDG Dose (RRFD) Cohort: Cohort I: Each participant (5 participants with bone tumor and 3 participants with lung tumor) underwent a CT simulation, then received a single injection of 15 mCi of FDG then underwent back-to-back RefleXion PET Imaging-Only session and third-party diagnostic PET/CT device. Each participant was then followed up at 72±24 hours after the imaging-only session.
- Cohort II: Delivery Emulation Cohort: Cohort II: The RRFD was determined in Cohort 1 as 15 mCi, after which enrollment began for Cohort II. In Cohort II each participant, (4 with bone tumor and 5 with lung tumor), underwent RefleXion PET image only sessions at three different timepoints. Each participant received a FDG injection of 15 mCi, prior to each image acquisition timepoint:
  The timepoints were as follows:
  1. At the time of enrollment: RefleXion PET image-only
  2: At SBRT First Fraction (Standard of Care): RefleXion PET Prescan #1
  3: At SBRT Last Fraction (Standard of Care): RefleXion PET Prescan #2 plus a Third-party PET/Scan.
  The participants were then followed-up at 72 ± 24 hours after final FDG injection.
Period: Overall Study
Arm/Group | Cohort I: Recommended RefleXion FDG Dose (RRFD) Cohort | Cohort II: Delivery Emulation Cohort
Started | 11 | 19
Enrolled (Received FDG Injection) | 8 | 9
Completed | 6 | 9
Not Completed | 5 | 10
Not completed — Screen Failure | 3 | 10
Not completed — Incomplete RMRS image session | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Cohort II: Delivery Emulation Cohort: Cohort II: The RRFD was determined in Cohort 1 as 15 mCi, aftter which enrollment began for Cohort II. In Cohort II each participant, (4 with bone tumor and 5 with lung tumor), underwent RefleXion PET image-only sessions at three different timepoints. Each participant received a FDG injection of 15 mCi, prior to each image acquisition:
  The timepoints were as follows:
  1. At the time of enrollment: RefleXion PET image-only
  2: At SBRT First Fraction (Standard of Care): RefleXion PET Prescan #1
  3: At SBRT Last Fraction (Standard of Care): RefleXion PET Prescan #2 plus a Third-party PET/Scan.
  The participants were then followed-up at 72 ± 24 hours after final FDG injection.
- Total: Total of all reporting groups
Arm/Group | Cohort I: Recommended RefleXion FDG Dose (RRFD) Cohort | Cohort II: Delivery Emulation Cohort | Total
Number analyzed (Participants) | 8 | 9 | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 6
  >=65 years | 5 | 6 | 11
Age, Continuous [Median (Full Range); unit: years]
  Cohort I & Cohort II | 68.01 [41 to 84] | 73.0 [57 to 87] | 70.5 [49 to 85.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 7 | 7 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 8 | 8 | 16
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 3 | 4
  White | 4 | 5 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Cohort I Recommended RefleXion FDG Dose (RRFD) to Enable the Use of BgRT Planning.
Description: The primary endpoint determined the number of cases that received the lowest FDG dose of 15 mCi, completed the RMRS image session and established an adequate target activity concentration to enable Biology guided Radiotherapy planning. The starting dose was 15mCi which was determined based upon preliminary physics studies done prior to this study. A FDG dose escalation to 20 mCi was not required.
Time Frame: During the RMRS imaging session
Population: The number of patients that received 15 mCi FDG dose and completed the RMRS image session.
Measure: Count of Participants; unit: Participants
Groups:
- Cohort I: Recommended RefleXion FDG Dose (RRFD): Cohort I: Each participant (5 participants with bone tumor and 3 participants with lung tumor) underwent a CT simulation, then received a single injection of 15 mCi of FDG then underwent back-to-back RefleXion PET Imaging-Only session and third-party diagnostic PET/CT device. Each participant was then followed up at 72±24 hours after the imaging-only session.
Arm/Group | Cohort I: Recommended RefleXion FDG Dose (RRFD)
Number analyzed (Participants) | 6
Participants | 6
Statistical Analysis 1: Comparison: Cohort I: Recommended RefleXion FDG Dose (RRFD); Statistical analysis of the primary endpoint is not applicable to Cohort I. A modified 3+3 design was utilized wherein meeting the activity level threshold, not dose-limiting toxicity, is the endpoint. The RRFD is primarily based upon the lower FDG dose level where 5 to 6 out of 6 subjects have an Activity Concentration greater than 5 kBq/ml."; Test type: Other — The modified 3+3 design with 6 patients at the 'Recommended RefleXion FDG Dose level' aims to ensure that the observed proportion of patients below activity threshold to be less than 33%. Probability of Observations at Most 1 of 6 below Activity Threshold True below activity rate 40% 30% 20% 10% Probability at most 1 of 6 patients below activity threshold 0.233 0.420 0.655 0.886; Statistical analysis of the primary endpoint is not applicable to Cohort I. A modified 3+3 design was utilized wherein meeting the activity level threshold, not dose-limiting toxicity, is the endpoint. The RRFD is primarily based upon the lower FDG dose level where 5 to 6 out of 6 subjects have an Activity Concentration greater than 5 kBq/ml."

2. Primary Outcome: Cohort II: Delivery Emulation
Description: The number of scans/fractions where the emulated BgRT dose distribution in a phantom was consistent with the BgRT treatment plan (i.e., 95% of DVH Delivered points for the BTZ and OAR fall within bounded DVH of the approved BgRT plan). There were 9 first fractions and 8 last fractions that were analyzed.
Time Frame: After SBRT First Fraction (standard of care) and after SBRT Last Fraction (standard of care)
Population: Cohort II - Emulated Delivery population evaluable scans
Measure: Count of Units; unit: Evaluable Fractions
Units Other Than Participants: Evaluable Fractions
Groups:
- Cohort II: Delivery Emulation Cohort: Cohort II: The RRFD was determined in Cohort 1 as 15 mCi, after which enrollment began for Cohort II. In Cohort II each participant, (4 with bone tumor and 5 with lung tumor), underwent RefleXion PET image-only sessions at three different timepoints. Each participant received a FDG injection of 15 mCi, prior to each image acquisition:
  The timepoints were as follows:
  1. At the time of enrollment: RefleXion PET image-only
  2: At SBRT First Fraction (Standard of Care): RefleXion PET Prescan #1
  3: At SBRT Last Fraction (Standard of Care): RefleXion PET Prescan #2 plus a Third-party PET/Scan.
  The participants were then followed-up at 72 ± 24 hours after final FDG injection.
Arm/Group | Cohort II: Delivery Emulation Cohort
Number analyzed (Participants) | 9
Number analyzed (Evaluable Fractions) | 17
Evaluable Fractions | 16

3. Secondary Outcome: Cohort I: Endpoint 1 Percent Agreement Between SI and AS for BgRT PET Imaging-only Session
Description: This endpoint evaluated percent of cases where there was an agreement between the site investigator SI and an Agreement Standard (AS) for the PET modeling localization decision. Six image comparisons were performed.
Time Frame: Immediately after RMRS imaging session
Population: The number of participants that received 15 mCi FDG dose injection and completed the RMRS image session.
Measure: Count of Participants; unit: Participants
Groups:
- Cohort I: Recommended RefleXion FDG Dose: Cohort I: Each participant (5 participants with bone tumor and 3 participants with lung tumor) underwent a CT simulation, then received a single injection of 15 mCi of FDG then underwent back-to-back RefleXion PET Imaging-Only session and third-party diagnostic PET/CT device. Each participant was then followed up at 72±24 hours after the imaging-only session.
Arm/Group | Cohort I: Recommended RefleXion FDG Dose
Number analyzed (Participants) | 6
Participants | 5

4. Secondary Outcome: Cohort I Endpoint 2: Percent of Cases X1 PET vs. Third-party Diagnostic PET/CT Image Comparison
Description: This endpoint evaluated Percent of cases where there was concordance of the positive "plan proceed" decision between the BgRT PET Imaging-only session and a third-party diagnostic PET/CT.
Time Frame: Immediately after RMRS imaging session
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort I: Recommended RefleXion FDG Dose
Number analyzed (Participants) | 6
Participants | 5

5. Secondary Outcome: Cohort I Endpoint 3: Biology Guided Radiotherapy (BgRT) Plan Generation
Description: Secondary Endpoint 3 evaluated the percent of cases where X1 PET images generated an Acceptable BgRT plan.
Time Frame: Immediately after RMRS imaging session
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort I: Recommended RefleXion FDG Dose
Number analyzed (Participants) | 6
Participants | 4

6. Secondary Outcome: Cohort I Endpoint 4: Percent of Cases Where the Intended Dose Distribution of BgRT Plan Was Achieved in the Physical Phantom.
Description: Secondary Endpoint 4 determined the percent of cases where the generated BgRT plan achieved acceptable quality assurance metrics in a physical phantom.
Time Frame: Immediately after RMRS imaging session
Measure: Count of Participants; unit: Participants
Groups:
- Cohort I: RRFD Cohort: Cohort I: Each participant (5 participants with bone tumor and 3 participants with lung tumor) underwent a CT simulation, then received a single injection of 15 mCi of FDG then underwent back-to-back RefleXion PET Imaging-Only session and third-party diagnostic PET/CT device. Each participant was then followed up at 72±24 hours after the imaging-only session.
Arm/Group | Cohort I: RRFD Cohort
Number analyzed (Participants) | 6
Participants | 6

7. Secondary Outcome: Cohort II Endpoint 1 Percent of Fractions With Concordance Between Physical and Digital Phantoms
Description: Number of fractions where there is concordance between the physical and digital phantoms of emulated BgRT delivery derived from human subject PET emissions. Concordance is defined as a standard gamma index with a goal that 90% of pixels meet the 3mm/3% deviation standard.
Time Frame: Assessed after SBRT First Fraction (standard of care) and after SBRT Last Fraction (standard of care), reported after SBRT Last Fraction.
Population: 17 scans for nine (9) subjects were used to measure the percent of fraction concordance between physical and digital phantoms of emulated BgRT delivery
Measure: Count of Units; unit: Fractions
Units Other Than Participants: Fractions
Arm/Group | Cohort II: Delivery Emulation Cohort
Number analyzed (Participants) | 9
Number analyzed (Fractions) | 17
Fractions | 17

8. Secondary Outcome: Cohort II Endpoint 2 Localization Decision
Description: Number of Pre-scan images where there is agreement between a site investigator and the agreement standard for the BgRT PET PreScan localization decision (overall percent agreement). Positive percent agreement and negative percent agreement will also be reported.
Time Frame: Assessed After PET Pre-Scan 1 and after PET Pre-Scan 2, reported after PET Pre-Scan 2.
Population: Cohort II Inter-observer agreement for Localization decision on RMRS PET Pre-Scan image
Measure: Count of Units; unit: PET Pre-Scan Image
Units Other Than Participants: PET Pre-Scan Image
Groups:
- Cohort II: Delivery Emulation Cohort: Cohort II: The RRFD was determined in Cohort I as FDG dose of 15 mCi. Following this Cohort II enrollment began.
  Each participant, 4 participants with bone tumor and 5 participants with lung tumor, underwent RefleXion PET image only sessions at three different timepoints. Prior to each the image collection the participant received a single dose injection of 15 mCi of FDG.
  1. At the time of enrollment: RefleXion PET image-only
  2: At SBRT First Fraction (Standard of Care): RefleXion PET Prescan #1
  3: At SBRT Last Fraction (Standard of Care): RefleXion PET Prescan #2 plus a Third-party PET/Scan.
  The subject was then followed-up at 72 ± 24 hours after final FDG injection.
Arm/Group | Cohort II: Delivery Emulation Cohort
Number analyzed (Participants) | 9
Number analyzed (PET Pre-Scan Image) | 18
PET Pre-Scan Image | 13

9. Secondary Outcome: Cohort II Endpoint 3 Image Concordance (Cohort II)
Description: Number of Scans where there is concordance of a positive localization decision between the short-duration PET PreScan and a third-party diagnostic PET/CT scan (positive percent agreement). Overall percent agreement and negative percent agreement will also be reported.
Time Frame: Assessed after Last fraction Imaging-only PET scan and Third-party PET/CT scan and reported after Third-party PET/CT scan.
Population: Comparison of short-duration PET CRR01 vs. Third-party Pet/CT
Measure: Count of Units; unit: Scans
Units Other Than Participants: Scans
Groups:
- Cohort II: Emulated Delivery Cohort: Cohort II: The RRFD was determined in Cohort 1 as 15 mCi, aftter which enrollment began for Cohort II. In Cohort II each participant, (4 with bone tumor and 5 with lung tumor), underwent RefleXion PET image-only sessions at three different timepoints. Each participant received a FDG injection of 15 mCi, prior to each image acquisition:
  The timepoints were as follows:
  1. At the time of enrollment: RefleXion PET image-only
  2: At SBRT First Fraction (Standard of Care): RefleXion PET Prescan #1
  3: At SBRT Last Fraction (Standard of Care): RefleXion PET Prescan #2 plus a Third-party PET/Scan.
  The participants were then followed-up at 72 ± 24 hours after final FDG injection.
Arm/Group | Cohort II: Emulated Delivery Cohort
Number analyzed (Participants) | 9
Number analyzed (Scans) | 7
Scans
  Positive Agreement | 7
  Overall agreement | 7

10. Secondary Outcome: Cohort II Endpoint 4 Toxicity Related to FDG Administrations
Description: Number of Participants who experienced AEs related to bladder and bone marrow assessed by complete blood count, urinalysis and AEs specific to bladder and bone marrow determined by Common Terminology Criteria for Adverse Events (CTCAE) v5 at 72±24 hours after final FDG injection.
Time Frame: Assessed at 72±24 hours after final FDG injection
Population: TEAE specific to Bladder or Bone Marrow
Measure: Number; unit: participants
Arm/Group | Cohort II: Emulated Delivery Cohort
Number analyzed (Participants) | 9
participants | 0

11. Secondary Outcome: Cohort II Endpoint 5 Workflow Characterization
Description: Workflow characterization by
  1. Number of participants with PET imaging-Only scans at RRFD that meet the Activity Concentration (AC) threshold for BgRT.
  2. Number of participants with PET imaging-Only scans that generate an acceptable BgRT plans.
  3. Number of participants with approved BgRT plans that Passed Physics Quality Assurance.
Time Frame: a. Immediately after RMRS imaging-Only sessions b. After acceptable BgRT plan generation c. During BgRT physics Quality Assurance
Population: PET imaging-Only sessions at RRFD that meets BTZ activation concentration threshold for BgRT (5 kBq/ml)
Measure: Count of Participants; unit: Participants
Groups:
- Cohort I - RRFD Cohort: Cohort I: All Participants, 5 participants with bone tumor and 3 participants with lung tumor, underwent CT simulations, received single injection of 15 mCi of FDG, underwent back-to-back RefleXion PET Imaging-Only session and third-party diagnostic PET/CT device and was followed up at 72±24 hours.
- Combined Cohort I + Cohort II: Combined Cohort I (RRFD Cohort) and Cohort II (Emulated Delivery Cohort) to characterize RefleXion system functioning
Arm/Group | Cohort I - RRFD Cohort | Cohort II: Delivery Emulation Cohort | Combined Cohort I + Cohort II
Number analyzed (Participants) | 6 | 9 | 15
Participants
  Number of participants with PET imaging-Only scans at RRFD meeting the AC threshold for BgRT. | 6 | 9 | 15
  b. Number of participants PET imaging sessions which lead to acceptable BgRT plans. | 4 | 9 | 13
  c. Number of participants approved BgRT plans that go on to pass physics quality assurance: number analyzed (Participants) | 4 | 9 | 13
  c. Number of participants approved BgRT plans that go on to pass physics quality assurance | 4 | 9 | 13

12. Secondary Outcome: Cohort II Endpoint 5d Workflow Characterization: PET Evaluations That Elicited a "Pass" Signal
Description: Number of PET Pre-Scans on the Day of Fraction Delivery that Elicited a "Pass" Signal Fraction Delivery.
Time Frame: Assessed after PET Pre-Scan 1 prior to First Fraction delivery and after PET Pre-Scan 2 prior to Last Fraction delivery, reported after PET Pre-Scan 2 prior to Last Fraction.
Population: Cohort II (Emulated Delivery Cohort)
Measure: Count of Units; unit: Scans
Units Other Than Participants: Scans
Arm/Group | Cohort II: Emulated Delivery Cohort
Number analyzed (Participants) | 9
Number analyzed (Scans) | 18
Scans | 17

ADVERSE EVENTS:
Time Frame: Cohort I -RRFD: AEs were collected starting at the time of injection of FDG and assessed at 72±24 hours after the end of Imaging-only session. Cohort II -Emulated Delivery: AEs were collected starting at time of first FDG injection and assessed at 72±24 hours after the final FDG injection.
Description: Any deaths, SAE, and other adverse events that started at the time of first FDG injection or 72±24 hours after the last FDG injection were collected in this study.
Groups:
- Cohort I: Recommended RefleXion FDG Dose (RRFD) Cohort: Cohort I: All Participants, 5 participants with bone tumor and 3 participants with lung tumor, underwent CT simulations, received single injection of 15 mCi of FDG, underwent back-to-back RefleXion PET Imaging-Only session and third-party diagnostic PET/CT device and was followed up at 72±24 hours.
Arm/Group | Cohort I: Recommended RefleXion FDG Dose (RRFD) Cohort | Cohort II: Delivery Emulation Cohort
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/9
Other Adverse Events (participants affected / at risk) | 5/8 | 5/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort I: Recommended RefleXion FDG Dose (RRFD) Cohort (N=8) | Cohort II: Delivery Emulation Cohort (N=9)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (2) — Shoulder pain
Back Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Oral Dysthesia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) — Decreased Appetite
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Somolence (Nervous system disorders) | 1 (1) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Creatinine Increased (Investigations) | 0 (0) | 1 (1) — Blood Creatinine Increase
Fatigue (General disorders) | 0 (0) | 2 (2)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Platelet count decrease (Investigations) | 0 (0) | 1 (1)
WBC decreased (Investigations) | 0 (0) | 1 (1)
Prostatic Obstruction (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Anemia (General disorders) | 0 (0) | 1 (1)
Lymphocyte count decrease (Investigations) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-23): https://cdn.clinicaltrials.gov/large-docs/47/NCT04788147/Prot_SAP_001.pdf